CLINICAL TRIAL: NCT05424874
Title: Clinical Validation of NAVOY® Acute Kidney Injury in Swedish ICU Patients
Acronym: ExTRACT
Status: Completed | Type: Observational
Sponsor: AlgoDx (Industry)
Responsible Party: Sponsor
Other Study IDs: AKI-SE-02
Record Dates: First submitted 2022-06-02; First posted 2022-06-21 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the performance of the prediction algorithm NAVOY® AKI in a Swedish adult ICU patient population versus fulfilment of KDIGO diagnostic criteria.

ELIGIBILITY:
Inclusion Criteria:

* The study will only include the subjects from the SEP-SE-02 study population. (NCT04570618)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult ICU patient population
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Prediction performance of NAVOY® AKI | Data from ICU stay between December 2020 to October 2021.
  The sensitivity, specificity, and accuracy will be calculated comparing the algorithm's predictions with the true AKI outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Sjövall, MD PhD, Principal Investigator — Skånes Universitetssjukhus
Locations (1):
- Intensiv- och perioperativ vård, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No